CLINICAL TRIAL: NCT07139665
Title: Investigation of Subacromial Space, Shoulder Pain, and Shoulder Disability Levels in Chronic Stroke Patients
Brief Title: Subacromial Space in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Büşra Seçkinoğulları Korkusuz, Principal Investigator, Ankara University
Other Study IDs: bbff9d0fc1ae4783
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Subacromial Space; Shoulder Pain; Shoulder Disability Levels
MeSH Terms: conditions — Stroke; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Stroke Patiens

SUMMARY:
This study aims to examine the subacromial space, shoulder pain, and shoulder disability in chronic stroke patients. A total of 60 chronic stroke patients aged 40-65 with similar demographic characteristics are planned to be included in this study. Participants will be selected voluntarily from among chronic stroke patients presenting for routine examination and follow-up at the Neurology Outpatient Clinic of Başkent University Hospital and meeting the appropriate inclusion criteria. Detailed demographic information (age, gender, stroke duration, affected side, etc.) will be recorded for all individuals included in the study.

DETAILED DESCRIPTION:
During the clinical assessment process, the subacromial space distance between the hemiplegic (affected) and healthy sides of the participants will be compared, and shoulder pain levels and shoulder disability levels will be examined. In this context, the subacromial space distance in the shoulder joint will be measured objectively using ultrasonography according to standard protocols. The severity of shoulder pain experienced by participants will be assessed subjectively using a Visual Analog Scale (VAS). Shoulder-related functional limitations and disability levels will be determined using a validated questionnaire, such as the Shoulder Pain and Disability Index (SPADI). Based on the data obtained, the relationships between subacromial distance, shoulder pain, and shoulder disability levels will be statistically analyzed. To ensure the statistical power of the study, a sample size target of 85% will be calculated, and additional individuals will be included if necessary to reach the specified sample size.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40 and 65.
* Scoring 21 or higher on the Montreal Cognitive Assessment Scale (MoCA).
* Being diagnosed with an ischemic or hemorrhagic stroke by a neurologist and having experienced the stroke for at least 6 months (chronic stroke).
* Scoring between 0 and 3 on the Modified Rankin Score.
* Volunteering to participate in the study

Exclusion Criteria:

* Difficulty with verbal communication (severe aphasia, cognitive impairment, etc.) that would prevent participation in the study and understanding the test instructions.
* Severe visual or hearing impairment that would affect test administration or safety.
* Having another neurological condition (e.g., Parkinson's disease, Multiple Sclerosis, severe peripheral neuropathy) other than stroke that could affect shoulder function or pain.
* Having a history of shoulder surgery before or after stroke, known rotator cuff tear, shoulder dislocation, severe degenerative joint disease (osteoarthritis), or inflammatory rheumatic disease (e.g., rheumatoid arthritis).
* Congestive heart failure, uncontrolled hypertension, or other serious cardiopulmonary disease that would preclude physical assessment or have exercise/positioning limitations.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Evaluation | Baseline
  In this study, ultrasonography will be used to objectively evaluate the subacromial space distance in the shoulder joint in chronic stroke patients.
Shoulder Pain and Disability Index | Baseline
  In this study, the Shoulder Pain and Disability Index will be used to subjectively assess participants' shoulder pain severity and shoulder-related functional limitations. The Shoulder Pain and Disability Index is a widely used, reliable, and valid self-report questionnaire for measuring pain and functional disability in individuals with shoulder problems.
Visual Analog Scale | Baseline
  The Visual Analog Scale is one of the pain rating scales frequently used in epidemiological and clinical studies to measure the intensity or frequency of various symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Ali Mert ÖZCAN, MSc, Study Chair — Baskent University; Ayşenur ÖZCAN, MSc, Study Chair — Çankırı Karatekin University; Sevgi İkbali Afşar, Prof. Dr., Study Chair — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tao W, Fu Y, Hai-Xin S, Yan D, Jian-Hua L. The application of sonography in shoulder pain evaluation and injection treatment after stroke: a systematic review. J Phys Ther Sci. 2015 Sep;27(9):3007-10. doi: 10.1589/jpts.27.3007. Epub 2015 Sep 30. PMID 26504346
- [Result] Seitz AL, Michener LA. Ultrasonographic measures of subacromial space in patients with rotator cuff disease: A systematic review. J Clin Ultrasound. 2011 Mar-Apr;39(3):146-54. doi: 10.1002/jcu.20783. Epub 2010 Dec 28. PMID 21387327
- [Result] Breckenridge JD, McAuley JH. Shoulder Pain and Disability Index (SPADI). J Physiother. 2011;57(3):197. doi: 10.1016/S1836-9553(11)70045-5. PMID 21843839